CLINICAL TRIAL: NCT00004825
Title: Short Term Study of Recombinant Human Insulin-like Growth Factor I in Children With Hyperinsulinism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Collaborators: Children's Hospital of Philadelphia (Other)
Purpose: Treatment
Other Study IDs: 199/13283; CHP-FDR001181-ST
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1998-07

CONDITIONS: Hyperinsulinism
Keywords: endocrine disorders; hyperinsulinism; rare disease
MeSH Terms: conditions — Hyperinsulinism; Endocrine System Diseases; Rare Diseases | interventions — Insulin-Like Growth Factor I

INTERVENTIONS:
Drug: recombinant human insulin-like growth factor I

SUMMARY:
OBJECTIVES: I. Confirm the inhibitory effect of recombinant human insulin-like growth factor I (IGF-I) on insulin secretion in children with hyperinsulinism.

II. Define the effects of short term IGF-I therapy on postprandial blood sugar levels in this patient population.

III. Characterize the effects of short term IGF-I therapy on fasting behavior, and other insulin dependent parameters, in this patient population.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Octreotide and/or diazoxide are discontinued on day 1, and fasting blood glucose is monitored. Patients receive test meals of Sustacal on days 3 and 4 and are assessed for insulin response.

Beginning on day 5, patients are given recombinant human insulin-like growth factor I subcutaneously every 12 hours for a total of 3 doses. The first dose (on day 5) is given 30 minutes before a Sustacal challenge, the second dose is followed by a bedtime snack, and the third dose (on day 6) is followed by a supervised fast.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Diagnosis of hyperinsulinism (i.e. evidence of fasting hypoglycemia with inadequate suppression of insulin, normal pituitary and adrenal function, and increased insulin action)

Suboptimal control of blood sugar (i.e. inability to fast at least 10 hours with a blood sugar of 60 mg/dL or greater)

No suspected insulinoma

Must be currently managed on a regimen of diazoxide, octreotide and/or frequent feedings to control hypoglycemia

--Prior/Concurrent Therapy--

See Disease Characteristics

--Patient Characteristics--

Hematopoietic: No anemia or other concerns of blood volume depletion

Renal: No renal dysfunction

Other:

* No known malignancy
* No other major medical conditions

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10
Dates: Start 1998-05; Study Completion 1998-05

CONTACTS AND LOCATIONS:
Overall Officials: Pinchas Cohen, Study Chair — Children's Hospital of Philadelphia